CLINICAL TRIAL: NCT05039021
Title: A Prospective, Single-Arm Multi-Center Study of the HARMONIC® 1100 Shears and Generator G11 in Pediatric Surgical Procedures (General) and Adult Surgical Procedures (General, Gynecological, Urological, and Thoracic)
Brief Title: A Prospective, Single-Arm Multi-Center Study of the HARMONIC® 1100 Shears in Select Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENG_2020_06
Record Dates: First submitted 2021-08-05; First posted 2021-09-09 (Actual); Results first posted 2025-03-12 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Pediatric Procedures; Adult Hepato-pancreato-biliary (HPB) Procedures; Adult Lower Gastrointestinal Procedures; Adult Gastric Procedures; Adult Gynecological Procedures; Adult Urological Procedures; Adult Thoracic Procedures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Pediatric; adult (HPB, lower gastrointestinal, gastric, gynecological, urological, thoracic) (Experimental): Any pediatric or adult (hepato-pancreato-biliary, lower gastrointestinal, gastric, gynecological, urological, thoracic) procedures where the HARMONIC 1100 Shears is used for vessel transection according to instructions for use.
  Interventions: Device: HARMONIC 1100 Shears

INTERVENTIONS:
Device: HARMONIC 1100 Shears — HARMONIC 1100 Shears is used for vessel transection according to instructions for use.

SUMMARY:
This prospective, single-arm, multi-center study will collect clinical data in a post-market setting for the pediatric population (general surgical procedures) and adult population (general, gynecological, urological, and thoracic surgical procedures). Investigators will perform each procedure using the device in compliance with their standard surgical approach and the HARMONIC 1100 Shears and Generator G11 instructions for use.

ELIGIBILITY:
Inclusion Criteria:

Pediatric population:

1. Non-emergent procedure (general) where at least one vessel is planned to be transected by the HARMONIC 1100 Shears per the IFU;
2. Less than 18 years of age at the time of procedure; and
3. The subject's parent/legal guardian must be willing to give permission for the subject to participate in the study and provide written informed consent for the subject. In addition, assent must be obtained from pediatric subjects who possess the intellectual and emotional ability to comprehend the concepts involved in the study. If the pediatric subject is not able to provide assent (due to age, maturity and/or inability to intellectually and/or emotionally comprehend the study), the parent/legal guardian's written informed consent for the subject will be acceptable for the subject to be included in the study.

Adult population:

1. Elective procedure (general, gynecological, urological, or thoracic) where at least one vessel is planned to be transected by the HARMONIC 1100 Shears per the IFU;
2. Willingness to give consent and comply with all study-related evaluations and visit schedule; and
3. At least 18 years of age.

Exclusion Criteria:

Preoperative

1. Physical or psychological condition which would impair study participation;
2. Female subjects, of childbearing age, who are pregnant; or
3. Enrollment in a concurrent interventional clinical study that could impact the study endpoints.

Intraoperative

1. The HARMONIC 1100 Shears were not attempted to be used for at least one single vessel transection during the surgical procedure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2024-02-04 (Actual); Study Completion 2024-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ethicon Endo-Surgery Clinical Trial, Study Director — Ethicon Endo-Surgery; Troy Markel, MD, Principal Investigator — Riley Hospital for Children at Indiana University Health; Attila Nakeeb, MD, Principal Investigator — IU Health University Hospital; Moishe Liberman, MD, Principal Investigator — Centre Hospitalier de l'Universite de Montreal
Locations (7):
- United States (4):
  - Baptist Health, Jacksonville, Florida
  - Indiana University, Indianapolis, Indiana
  - IU Health University Hospital, Indianapolis, Indiana
  - Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana
- Canada (2):
  - Centre Hospitalier de l'Universite de Montreal, Montreal
  - Toronto General Hospital, Toronto
- Western General Hospital, Edinburgh, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- HARMONIC 1100 Shears: HARMONIC 1100 Shears was used per the Instructions for use (IFUs) in pediatric surgical procedures (general) or adult surgical procedures (general, gynecological, urological, and thoracic) where at least one single vessel was transected.
Period: Overall Study
Arm/Group | HARMONIC 1100 Shears
Started | 265
Completed | 261
Not Completed | 4
Not completed — Death | 1
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | HARMONIC 1100 Shears
Number analyzed (Participants) | 265
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.73 (22.793)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 158
  Male | 107
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 224
  Unknown or Not Reported | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 29
  White | 213
  More than one race | 0
  Unknown or Not Reported | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Vessels Transected With Less Than or Equal to (<=) Grade 3 Hemostasis Based on Hemostasis Grading Scale
Description: Number of vessels transected with <= Grade 3 hemostasis based on hemostasis grading scale were reported. A 4-point grading scale was used to assess hemostasis in blood vessels. Grade 1: no bleeding at transection site; Grade 2: minor bleeding at transection site, no intervention needed; Grade 3: minor bleeding at transection site, mild intervention needed, use of compression, monopolar device and/or touch-ups with HARMONIC 1100 Shears; or Grade 4: significant bleeding (example, pulsatile blood flow, venous pooling) requiring intervention such as extensive coagulation or use of additional hemostatic measures (example, hemoclips, staples, sutures, fibrin sealants, other advanced energy products).
Time Frame: On the day of transection (Day 0)
Population: Full analysis set included participants in whom the HARMONIC 1100 Shears was utilized during the surgical procedure to transect at least one vessel. Here, "Overall number of units analyzed" signifies total number of vessels transected and analyzed for this outcome measure.
Measure: Count of Units; unit: Vessels transected
Units Other Than Participants: Vessels transected
Arm/Group | HARMONIC 1100 Shears
Number analyzed (Participants) | 265
Number analyzed (Vessels transected) | 489
Vessels transected | 484

2. Primary Outcome: Number of Participants With Device-related Adverse Events (AEs)
Description: Number of participants with device-related AEs were reported. Device-related AEs were those AEs identified as having a relationship of possibly, probably, or causally with the study device. Possible refers to the relationship with the use of the device is weak but cannot be ruled out completely; Probable refers to the relationship with the use of the device seems relevant and/or the event cannot reasonably be explained by another cause, but additional information may be obtained; Causal relationship refers to the event is associated with the device or with procedures beyond reasonable doubt.
Time Frame: From Day 0 up to post-procedure follow up visit (up to 28 days)
Population: Safety analysis set included participants in whom the HARMONIC 1100 Shears was utilized during the surgical procedure to transect at least one vessel.
Measure: Count of Participants; unit: Participants
Arm/Group | HARMONIC 1100 Shears
Number analyzed (Participants) | 265
Participants | 5

3. Secondary Outcome: Number of Vessels Transections With Diameter >5 to 7 mm With Less Than or Equal to (<=) Grade 3 Hemostasis Based on Hemostasis Grading Scale
Description: Number of vessels transected with diameter >5 to 7 mm with <= Grade 3 hemostasis based on hemostasis grading scale were reported. A 4-point grading scale was used to assess hemostasis in blood vessels. Grade 1: no bleeding at transection site; Grade 2: minor bleeding at transection site, no intervention needed; Grade 3: minor bleeding at transection site, mild intervention needed, use of compression, monopolar device and/or touch-ups with HARMONIC 1100 Shears; or Grade 4: significant bleeding (example, pulsatile blood flow, venous pooling) requiring intervention such as extensive coagulation or use of additional hemostatic measures (example, hemoclips, staples, sutures, fibrin sealants, other advanced energy products).
Time Frame: On the day of transection (Day 0)
Population: as for outcome 1
Measure: Count of Units; unit: Vessels transected
Units Other Than Participants: Vessels transected
Arm/Group | HARMONIC 1100 Shears
Number analyzed (Participants) | 265
Number analyzed (Vessels transected) | 489
Vessels transected | 174

4. Secondary Outcome: Number of Participants Using HARMONIC 1100 Shears For Sealing and Transection of Lymphatic Vessels as Assessed by Surgeon Satisfaction Scale Score
Description: Number of participants using HARMONIC 1100 Shears for sealing and transection of lymphatic vessels as assessed by Surgeon Satisfaction Scale Score were reported. Surgeon satisfaction scale score is a 5-point scale (very dissatisfied, dissatisfied, neither satisfied or dissatisfied, satisfied, or very satisfied) where surgeon rated the use of the device for sealing and transection of lymphatic vessel by HARMONIC 1100 Shears.
Time Frame: On the day of transection (Day 0)
Population: Analysis population included participants in FAS with sealing and transection of lymphatic vessels by HARMONIC 1100 Shears.
Measure: Count of Participants; unit: Participants
Arm/Group | HARMONIC 1100 Shears
Number analyzed (Participants) | 104
Participants
  Very Satisfied | 76
  Satisfied | 25
  Neither Satisfied or Dissatisfied | 0
  Dissatisfied | 0
  Very Dissatisfied | 3

5. Secondary Outcome: Number of Vessels Transected With Hemostasis (Grade 1 to 4) Based on Hemostasis Grading Scale
Description: Number of vessels transected with hemostasis (Grade 1 to 4) based on hemostasis grading scale was reported. A 4-point grading scale was used to assess hemostasis in blood vessels. Grade 1: no bleeding at transection site; Grade 2: minor bleeding at transection site, no intervention needed; Grade 3: minor bleeding at transection site, mild intervention needed, use of compression, monopolar device and/or touch-ups with HARMONIC 1100 Shears; or Grade 4: significant bleeding (example, pulsatile blood flow, venous pooling) requiring intervention such as extensive coagulation or use of additional hemostatic measures (example, hemoclips, staples, sutures, fibrin sealants, other advanced energy products).
Time Frame: On the day of transection (Day 0)
Population: as for outcome 1
Measure: Count of Units; unit: Vessels transected
Units Other Than Participants: Vessels transected
Arm/Group | HARMONIC 1100 Shears
Number analyzed (Participants) | 265
Number analyzed (Vessels transected) | 489
Vessels transected
  Grade 1 | 475
  Grade 2 | 2
  Grade 3 | 7
  Grade 4 | 5

6. Secondary Outcome: Number of Grade 4 Vessel Transections Requiring Hemostasis Measures
Description: Number of Grade 4 vessel transections requiring hemostasis measures such as hemoclips, staples, sutures, fibrin sealants, adjunctive topical hemostats (except fibrin sealants), other advanced energy products and other products were reported. A 4-point grading scale was used to assess hemostasis in blood vessels. Grade 1: no bleeding at transection site; Grade 2: minor bleeding at transection site, no intervention needed; Grade 3: minor bleeding at transection site, mild intervention needed, use of compression, monopolar device and/or touch-ups with HARMONIC 1100 Shears; or Grade 4: significant bleeding (pulsatile blood flow, venous pooling) requiring intervention such as extensive coagulation or use of additional hemostatic measures (hemoclips, staples, sutures, fibrin sealants, adjunctive topical hemostats (except fibrin sealants), other advanced energy products). Since multiple responses were collected, sum of the data of each category exceeds the overall number of units analyzed.
Time Frame: On the day of transection (Day 0)
Population: Full analysis set included participants in whom the HARMONIC 1100 Shears was utilized during the surgical procedure to transect at least one vessel. Here, 'N' (overall number of participants analyzed) signifies number of participants evaluable for this outcome measure. Here, "Overall number of units analyzed" signifies Grade 4 vessels transections.
Measure: Count of Units; unit: Vessels transected
Units Other Than Participants: Vessels transected
Arm/Group | HARMONIC 1100 Shears
Number analyzed (Participants) | 4
Number analyzed (Vessels transected) | 5
Vessels transected
  Hemoclips | 4
  Staples | 1
  Sutures | 0
  Fibrin Sealants | 0
  Adjunctive Topical Hemostats (except Fibrin Sealants) | 1
  Other Advanced Energy Products | 1
  Other | 1

ADVERSE EVENTS:
Time Frame: From Day 0 up to post-procedure follow up visit (Up to 28 days)
Description: Safety analysis set included participants in whom the HARMONIC 1100 Shears was utilized during the surgical procedure to transect at least one vessel.
Arm/Group | HARMONIC 1100 Shears
All-Cause Mortality (participants affected / at risk) | 1/265
Serious Adverse Events (participants affected / at risk) | 16/265
Other Adverse Events (participants affected / at risk) | 69/265
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HARMONIC 1100 Shears (N=265)
Acute myocardial infarction (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Abdominal pain lower (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2
Empyema (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Post procedural pneumonia (Infections and infestations) | 1
Anastomotic complication (Injury, poisoning and procedural complications) | 1
Anastomotic leak (Injury, poisoning and procedural complications) | 1
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 1
Procedural nausea (Injury, poisoning and procedural complications) | 1
Procedural vomiting (Injury, poisoning and procedural complications) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1
Circulatory collapse (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HARMONIC 1100 Shears (N=265)
Anaemia (Blood and lymphatic system disorders) | 4
Blood loss anaemia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 7
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Abdominal tenderness (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 2
Epigastric discomfort (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 9
Odynophagia (Gastrointestinal disorders) | 2
Retching (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 3
Chest pain (General disorders) | 1
Hernia (General disorders) | 1
Pain (General disorders) | 8
Pyrexia (General disorders) | 3
Bronchitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Fungaemia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Postoperative wound infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 5
Anastomotic haemorrhage (Injury, poisoning and procedural complications) | 1
Confusion postoperative (Injury, poisoning and procedural complications) | 1
Incision site pain (Injury, poisoning and procedural complications) | 1
Incision site pruritus (Injury, poisoning and procedural complications) | 1
Incision site vesicles (Injury, poisoning and procedural complications) | 1
Penis injury (Injury, poisoning and procedural complications) | 1
Post procedural discomfort (Injury, poisoning and procedural complications) | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 1
Procedural nausea (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 5
Splenic injury (Injury, poisoning and procedural complications) | 1
Wound complication (Injury, poisoning and procedural complications) | 3
Wound haemorrhage (Injury, poisoning and procedural complications) | 1
Wound secretion (Injury, poisoning and procedural complications) | 3
Aspiration pleural cavity (Investigations) | 1
Blood glucose increased (Investigations) | 1
Creatinine renal clearance decreased (Investigations) | 1
Glomerular filtration rate decreased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Oxygen saturation decreased (Investigations) | 2
Urine output decreased (Investigations) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 1
Bladder discomfort (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Breast pain (Reproductive system and breast disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 3
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 1
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1
Arterial haemorrhage (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 1
Hot flush (Vascular disorders) | 1
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Draft abstracts, manuscripts, and materials for presentation at scientific meetings must be sent to the sponsor at least 60 working days prior to abstract or other relevant submission deadlines. Authorship of publications resulting from this study was based on generally accepted criteria for major medical journals.

DOCUMENTS (2):
  • Study Protocol (2023-05-17): https://cdn.clinicaltrials.gov/large-docs/21/NCT05039021/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-06): https://cdn.clinicaltrials.gov/large-docs/21/NCT05039021/SAP_001.pdf